CLINICAL TRIAL: NCT07157462
Title: Investigation of the Effects of a Multispecies Probiotic Formulation on Perennial Allergic Rhinitis
Acronym: AllerGo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Winclove B.V. (Industry)
Collaborators: Alyatec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIN-001
Record Dates: First submitted 2025-08-21; First posted 2025-09-05 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Multispecies probiotic; House dust mite allergy; cat and dog allergy
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Dust Mite Allergy | interventions — Lacteol; Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Participants receive a multispecies probiotic formulation for oral use
  Interventions: Dietary Supplement: Multi-species probiotic powder for oral solution. Dietary supplement containing six bacterial strains (Lactobacillus and Bifidobacterium species)
- Placebo (Placebo Comparator): The participants receive a placebo for oral use, comparable in appearance and smell as the probiotic formulation
  Interventions: Dietary Supplement: Placebo Powder for Oral Solution

INTERVENTIONS:
Dietary Supplement: Multi-species probiotic powder for oral solution. Dietary supplement containing six bacterial strains (Lactobacillus and Bifidobacterium species) — The probiotic powder is provided in sachets. The Participants dissolve the powder in water and ingest twice daily for 12 weeks.
  Arms: Probiotic
Dietary Supplement: Placebo Powder for Oral Solution — The placebo powder is provided in sachets. The Participants dissolve the powder in water and ingest twice daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if a probiotic formulation consisting of multiple bacterial strains has a positive effect on the quality of life of participants with chronic perennial allergic rhinitis symptoms. The researchers will also study whether the probiotic formulation influences the symptoms of allergic rhinitis. Participants with allergies to house dust mite, cats and/or dogs will be included in the study.

The main questions it aims to answer are:

Does the probiotic formulation have an impact of the quality of life of the participants? Does the probiotic formaluation have an effect on the severity of the symptoms of allergic rhinitis? Are there differences in the effects depending on the allergies the participants have?

Researchers will compare the probiotic formulation to a placebo (a substance that contains no probiotic bacteria but looks, smells, and tastes the same) to see if the probiotic formulation improves the quality of life of participants with chronic allergic rhinitis. In addition, also a GI symptom questionnaire will be filled in by the participants weekly

Participants will visit the clinic for the screening, and at the start, and at the end of the intervention for checkups and sampling. During the intervention they will take the probiotic formulation or a placebo twice every day for 12 weeks. They will keep a diary of their symptoms and note whenever they use anti-histamines and every two weeks they will fill in a questionnaire about their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Willing and able to provide informed consent in French
* Persistent perennial allergic rhinitis induced by a least one perennial allergen in the last two years.
* Positive skin prick test ≥5 mm for any of the following allergens: cat, dog and mites
* Mean global score of miniRQLQ ≥ 2
* TSS score of at least 7
* Willing to discontinue consumption of fermented foods, probiotics (e.g., yogurts with live, active cultures or supplements), prebiotics or immune-enhancing supplements (e.g., Echinacea or fish oil).
* Agreement on not starting new medication during the intervention (rescue medication excepted)
* Women of childbearing potential with a negative pregnancy test throughout the study period and highly effective contraception: oral contraceptives, condom with spermicide, intrauterine device, bilateral tubal ligation, vasectomized partner

Exclusion Criteria:

* Non-allergic rhinitis
* Use of any prohibited medication (any systemic corticosteroids, androgens such as testosterone, or high doses of anti-inflammatory drugs: i.e., aspirin in doses 600 mg/d regularly) at the time of enrolment
* Use of other probiotics-containing and prebiotics-containing products during the intervention period and 4 weeks before study start
* Use of any antibiotics 6 weeks before randomization
* Nasal polyposis
* Currently enrolled in another intervention study (except observational studies)
* Critically or terminally ill or admitted to the ICU
* Had received chemotherapy or other immune-suppressing therapy within the previous year.
* Other conditions that according to the investigator might interfere with the evaluation of the study objectives
* Patients being treated for or had any of the following physician-diagnosed diseases or conditions: HIV; immune modulating diseases (autoimmune disease, hepatitis, cancer, etc.); kidney disease; pancreatitis; pulmonary disease; hepatic or biliary disease; or gastrointestinal diseases or conditions, such as diverticulitis, ulcerative colitis, Crohn's disease, Celiac disease, short bowel disease, ileostomy, or colostomy, but not including gastroesophageal reflux disease,
* Subjects with a low compliance rate (appreciated by the investigator) during the run-in period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the change in the global score of the mini-Rhinoconjunctivitis Quality of Life Questionnaire (mini-RQLQ) from baseline to week 12 of intervention | From baseline to 12 weeks of intervention
  An improvement on quality of life is considered clinically meaningful when improved with ≥0.7 points in global and domain-specific mini-RQLQ scores between intervention and placebo

SECONDARY OUTCOMES:
The impact of intervention in rhino conjunctivitis quality of life will be assessed by the changes in global and domain-specific mini-RQLQ scores from baseline to week 12 of intervention every two weeks. | Every two weeks from baseline to end of treatment at 12 weeks
The proportion of participants reporting a clinical relevant improvement on quality of life in global and domain-specific mini-RQLQ scores between intervention and placebo | From baseline to end of treatment at 12 weeks
  The proportion of participants reporting a clinical relevant improvement on quality of life will be assessed by the difference in proportion of participants achieving a clinically meaningful improvement (≥0.7 points) in global and domain-specific mini-RQLQ scores between intervention and placebo
The proportion of participants reporting a clinical relevant improvement on allergic rhinoconjuctivitis symptoms in global and domain-specific TSS scores between intervention and placebo | From baseline to end of treatment at 12 weeks
  The proportion of participants reporting a clinical relevant improvement on allergic rhinoconjuctivitis symptoms will be assessed by the difference in proportion of participants achieving a clinically meaningful improvement (≥20%) in global and domain-specific TSS scores between intervention and placebo
The impact of a multispecies probiotic formulation on allergic rhinoconjunctivitis severity will be assessed by the difference in TSS mean (global and per item) between intervention and placebo over 12 weeks. | From baseline to end of treatment at 12 weeks, daily
The impact of a multispecies probiotic formulation on allergic rhinoconjunctivitis severity with established perennial allergies will be assessed as the change in the global score of the TSS from baseline to week 12 of intervention. | From baseline to end of treatment at 12 weeks
Differences in TSS will be analysed in subgroups of participants based on type of allergy | From baseline to end of treatment at 12 weeks, daily
  Differences in TSS will be analysed in subgroups of participants based on type of allergy (HDM, HDM+Cat, HDM+Cat+Dog, Cat, Cat+Dog and Dog)
Differences in TSS will be analysed in subgroups of participants based on allergy pattern | From baseline to end of treatment at 12 weeks, daily
  Differences in TSS will be analysed in subgroups of participants based on different allergy pattern (perennial vs perennial with seasonal allergies)
Differences in TSS will be analysed in subgroups of participants based on baseline severity of TSS score | From baseline to end of treatment at 12 weeks, daily
  Differences in TSS will be analysed in subgroups of participants based on baseline severity as stratified by TSS scores as follows: 0-6 = mild, 7-12=moderate, 13-18 =moderate/severe, and 19-24= severe
Differences in mini-RQLQ will be analysed in subgroups of participants based on type of allergy | From baseline to end of treatment at 12 weeks, two weekly
  Differences in mini-RQLQ will be analysed in subgroups of participants based on type of allergy (HDM, HDM+Cat, HDM+Cat+Dog, Cat, Cat+Dog and Dog)
Differences in mini-RQLQ will be analysed in subgroups of participants based on allergy pattern | From baseline to end of treatment at 12 weeks, two weekly
  Differences in mini-RQLQ will be analysed in subgroups of participants based on on different allergy pattern (perennial vs perennial with seasonal allergies)
Differences in mini-RQLQ will be analysed in subgroups of participants based on baseline severity of mini-RQLQ | From baseline to end of treatment at 12 weeks, two weekly
  Differences in mini-RQLQ will be analysed in subgroups of participants based on baseline severity as stratified by mini-RQLQ as follows: 0-1.5, 1.5-2.5, 2.5-3.5, 3.5-4.5, >4.5
Change in immune modulatory biomarkers (cytokines and IgE) at baseline compared to 12 weeks of intervention versus placebo | From baseline to end of treatment at 12 weeks
Change in amount of blood cells at baseline compared to 12 weeks of intervention versus placebo | From baseline to end of treatment at 12 weeks
Change in ratio of blood cell at baseline compared to 12 weeks of intervention versus placebo | From baseline to end of treatment at 12 weeks
Change in rescue medication use (antihistamines) will be expressed as a percentage of the completed daily diary entries over the 12 weeks intervention period | From baseline to end of treatment
Reduction in gastro-intestinal complaints will be assessed using the GSRS questionnaire after 12 weeks intervention versus placebo and across weekly time points | From baseline to end of treatment at 12 weeks and weekly between those timepoints
Reduction in allergic symptoms other than rhinitis (eczema, food allergy and intolerance) using Non-rhinoconjunctivitis allergy Questionnaire over the 12 weeks intervention versus placebo | From baseline to end of treatment at 12 weeks
Change in fecal microbiome profile or metabolites production (e.a SCFA and bile acids) will be analyzed after 12 weeks intervention versus placebo | From baseline to end of treatment at 12 weeks

OTHER OUTCOMES:
Correlation between change from baseline in GSRS total score and changes in gut microbiome composition and fecal metabolite concentrations at Week 12 | From baseline to end of treatment at 12 weeks
  Associations between gastrointestinal symptom changes, as measured by the Gastrointestinal Symptom Rating Scale (GSRS; 15 items, 7-point Likert scale), and changes in gut microbiome composition and fecal metabolite concentrations will be explored. Microbiome profiling will be performed using 16S rRNA sequencing of stool samples, and metabolite analysis will include short-chain fatty acids (SCFAs), bile acids, and other metabolites identified through untargeted metabolomics. Correlation analyses (e.g., Spearman's rank correlation) and/or linear regression models will be applied. Additional multivariate or network analyses may be used to explore complex interaction patterns. These analyses are exploratory and hypothesis-generating; no formal adjustment for multiple testing will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Alina GHERASIM, MD, Principal Investigator — ALYATEC clinical center
Locations (1):
- ALYATEC clinical center, Strasbourg, Alyatec, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated and anonymized data will be analyzed and reported. The individual participant data are collected and managed by the contract research organization (CRO) and remain confidential. Data will be presented in summary form in scientific publications and regulatory submissions only.